CLINICAL TRIAL: NCT00758212
Title: Influenza Vaccination at a Reduced Dose of 1:10 Using Mesotherapy in HIV/AIDS Patients at the Hadassah AIDS Center, Jerusalem
Brief Title: Influenza Vaccination at a Reduced Dose Using Mesotherapy in HIV/AIDS Patients at the Hadassah AIDS Center, Jerusalem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Shlomo Maayan MD ; Director, Hadassah AIDS Center, Hadassah Medical organization
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: azw6gmHHMO-CTIL
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-09

CONDITIONS: Influenza; Acquired Immune Deficiency Syndrome; HIV Infections
Keywords: Influenza in Humans; Acquired Immune Deficiency Syndrome; Immunization, Active
MeSH Terms: conditions — Influenza, Human; Acquired Immunodeficiency Syndrome; HIV Infections; Motor Activity | interventions — Mesotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): The experimental group will consist of HIV/AIDS patients(approx.50) who volunteer to receive a reduced dose Influenza vaccine using mesotherapy as a mode of injecting the vaccine intradermally.
  Interventions: Biological: Mesotherapy

INTERVENTIONS:
Biological: Mesotherapy — The regular seasonal trivalent Influenza vaccine( Vaxigrip) will be diluted 1:10 in saline.The diluted vaccine will be given intra-dermally using Mesotherapy,namely multiple injections given at one time in the torso, back and axillae.
  Other Names: Vaxigrip Trivalent Influenza vaccine , diluted 1:10.

SUMMARY:
Influenza vaccination has proved it's effectiveness over many years of usage including HIV/AIDS patients who are immunocompromised. In those patients, however, a noted rise in HIV viral load which follows intramuscular injection of the vaccine is of unknown significance over the long run. Mesotherapy is a procedure developed and practiced in france by which a reduced and diluted amounts of antigens is being introduced by multiple intradermal injections over the torso and upper back. Mesotherapy is mainly used as a vehicle for introducing pain medicine and cosmetics.

DETAILED DESCRIPTION:
We will test the effectiveness of mesotherapy as a vehicle for influenza vaccination.We will use 1:10th of the amount of seasonal trivalent influenza vaccine in approx.50 HIV/AIDS patients.A control group of approx.50 matched patients for age ,treatment schedule and immune status will receive the regular injection of trivalent vaccine. We will follow patients clinically for symptoms compatible with seasonal influenza and for direct side effects of the vaccine.In addition we will measure anti influenza antibody in the two groups .Follow up will be for 6 months following vaccination.Anti influenza antibody will be measured at 1,3,6months using hemagglutination inhibition (HAI) test.

ELIGIBILITY:
Inclusion Criteria:

* Virologic diagnosis of HIV/AIDS.
* Any immune derangement is acceptable

Exclusion Criteria:

* Allergy to eggs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-01 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
anti influenza antibody using Hemagglutination inhibition | 1 , 3 , 6 months

SECONDARY OUTCOMES:
acceptability of influenza vaccination using mesotherapy | 1month

CONTACTS AND LOCATIONS:
Overall Officials: shlomo maayan, md, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah U. hospital, Jerusalem, Israel

REFERENCES:
- [Background] Lin JC, Nichol KL. Excess mortality due to pneumonia or influenza during influenza seasons among persons with acquired immunodeficiency syndrome. Arch Intern Med. 2001 Feb 12;161(3):441-6. doi: 10.1001/archinte.161.3.441. PMID 11176770
- [Background] Kenney RT, Frech SA, Muenz LR, Villar CP, Glenn GM. Dose sparing with intradermal injection of influenza vaccine. N Engl J Med. 2004 Nov 25;351(22):2295-301. doi: 10.1056/NEJMoa043540. Epub 2004 Nov 3. PMID 15525714